CLINICAL TRIAL: NCT03221296
Title: A Feasibility Study on the Effects of Vestibular Training as a Fall Prevention Strategy in the Elderly
Brief Title: Fall Prevention - Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Carmela Tartaglia, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-5055
Record Dates: First submitted 2017-07-07; First posted 2017-07-18 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer Dementia (AD); Vascular Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular Training (Intervention Group) (Experimental): For the actual intervention, participants will be asked to commit a total of approximately 20 minutes a day of vestibular exercise, divided into three separate sessions (i.e. three 7 minute sessions).
  These will include eye movement exercises, walking and balancing. Every 2 weeks, there will be a slight change to the exercises to increase difficulty. (i.e. balancing on one leg or walking with head turns)
  Interventions: Behavioral: Vestibular Training (Intervention Group)
- Usual Care (Control group) (No Intervention): Patients that are randomized to standard of care Control group will undergo Baseline and 12-week assessments including vestibular testing and questionnaires.

INTERVENTIONS:
Behavioral: Vestibular Training (Intervention Group) — Exercises three times daily, for up to approximately 20 minutes. Changes in functional status and physical status shall be measured at study onset and follow up.
  Arms: Vestibular Training (Intervention Group)

SUMMARY:
A feasibility study of a vestibular rehabilitation program in a sample of cognitively impaired clinical patients to guide future trials.

DETAILED DESCRIPTION:
This is a feasibility study to gather preliminary data on a vestibular rehabilitation program. All participants who visit UHN memory clinic with a diagnosis of mild/moderate cognitive impairment due to Alzheimer's or vascular disease or both and have had falls will be asked to participate. If agree to be contacted they will receive a consent form.

All agreeable participants shall be screened for vestibular impairment through the following tests: Dix-Hall pike test, Head Impulse Test, Head Shake test, test of Dynamic Visual Acuity. In addition, participants will complete the MoCA to assess cognitive functioning. A score lower than 15 will exclude the participant.

After determining the population who is eligible for this study and willing to participate, participants shall move to baseline assessment. At baseline, measurements of balance, gait, and dynamic visual acuity in addition to questionnaires about dizziness felt, confidence in performing activities without falling, depression and quality of life, shall be completed.

Immediately after baseline, participants will begin their treatment arm, depending on if they have been put in the vestibular group or control group. Participants in the vestibular arm will be taught vestibular exercises and asked to perform vestibular exercises for 3 sessions daily, 3-10 minutes/session. Participation in vestibular exercises shall be recorded via a log by their caregiver. During the 12 weeks, these diaries shall be kept with the participant caregiver. Caregivers shall be followed up bi-weekly to ensure that participants are completing the exercises, and logging their participation.

At the end of the 12 weeks, participants will be reassessed with the same measures from baseline in addition to the head impulse test and test of dynamic visual acuity. The investigators shall also administer a final questionnaire (Problematic Experiences of Therapy Scale) to see what may have prevented completion of therapy or caused issues.

Participants that are randomized to standard of care Control group will undergo Baseline and 12-week assessments including vestibular testing and questionnaires.

3-months after final assessments (6 months after start), all participants shall be contacted to see if there were any falls/near fall experiences.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people ages 65 and older
* English speaking
* Can log their participation or have a caregiver log on their behalf
* Mild/moderate dementia [(1) Alzheimer's disease, (2) small vessel vascular dementia not related to stroke and (3) mixed dementia of Alzheimer's or small vessel vascular not related to stroke] or mild/moderate cognitive impairment
* Vestibular Impairment

Exclusion Criteria:

* Neurological disease (e.g. seizures, stroke, hemorrhage, central nervous system tumor, multiple sclerosis)
* Being diagnosed with a psychiatric disorder (e.g. Major depression episode, post-traumatic stress disorder, generalized anxiety disorder, schizophrenia, bipolar disorder etc.)
* Those with a current inner ear infection
* Those with severe neck arthritis
* Those with Post-Concussion Syndrome
* Severe cognitive impairment as defined by a MoCA <15
* Following etiologies of dementia: Dementia due to Lewy bodies, Parkinson's disease, Huntington's Disease, Frontotemporal Dementia, Normal Pressure Hydrocephalous

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Number of falls/near fall experiences through the Falls Video Analysis Questionnaire (FVAQ) | 3 months and again 6 months after baseline
  Measured by comparing the test score change from baseline to follow up at 3 months and again at 6 months to determine if the therapy worked

SECONDARY OUTCOMES:
Change in levels of dizziness through the Dizziness Handicap Inventory (DHI) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Change in perceived level of confidence through the Activities Specific Balance Confidence Scale (ABC) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Change in quality of life through The Geriatric Depression Scale (GDS) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Cognitive status through the Montreal Cognitive Assessment (MoCA) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Change in physical functioning through the head impulse test (HIT) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Number of patients who can successfully complete Head Impulse Test (HIT) | 3 months
  Shall be measured by proportion of participants completing test (did not need to stop for any reason)
Number of patients who can successfully complete Head Shake Test (HST) | 3 months
  Shall be measured by proportion of participants completing test (did not need to stop for any reason)
Number of patients who can successfully complete Dynamic Gait Index (DGI) | 3 months
  Shall be measured by proportion of participants completing test (did not need to stop for any reason)
Number of patients who can successfully complete the test of dynamic visual acuity (DVA) | 3 months
  Shall be measured by proportion of participants completing test (did not need to stop for any reason)
Number of patients who can successfully complete the modified clinical test of sensory interaction on balance (mCTSIB) | 3 months
  Shall be measured by proportion of participants completing test (did not need to stop for any reason)
Completeness of questionnaires and which questions were: skipped, missed or difficult to understand for the Dizziness Handicap Inventory (DHI) | 3 months
  Shall be measured by percentage of test items completed
Completeness of questionnaires and which questions were: skipped, missed or difficult to understand for the Montreal Cognitive Assessment (MoCA) | 3 months
  Shall be measured by percentage of test items completed
Completeness of questionnaires and which questions were: skipped, missed or difficult to understand for the Quality of Life in Alzheimer's Disease (QOL-AD) | 3 months
  Shall be measured by percentage of test items completed
Completeness of questionnaires and which questions were: skipped, missed or difficult to understand for the World Health Organization Quality of Life - BREF (WHOQOL-BREF) | 3 months
  Shall be measured by percentage of test items completed
Completeness of questionnaires and which questions were: skipped, missed or difficult to understand for the Activities Specific Balance Confidence scale (ABC) | 3 months
  Shall be measured by percentage of test items completed
Completeness of questionnaires and which questions were: skipped, missed or difficult to understand for the Geriatric Depression Scale (GDS) | 3 months
  Shall be measured by percentage of test items completed
Number of patients who successfully adhered to the vestibular rehabilitation program through the Problematic Experiences of Therapy scale (PETs) | 3 months
  filled out by both, or either one of, the patient or caregiver
Attrition Rate | 3 months
  Will be measured as the percentage of those who reached follow-up compared to those who completed baseline
Number of patients willing to participate | 3 months
  Determined by the proportion of patients saying yes out of those contacted
Change in quality of life through The World Health Organization Quality of Life - BREF (WHOQOL-BREF) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Change in quality of life through The Quality of Life in Alzheimer's Disease (QOL-AD) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Change in physical functioning through the head shake test (HST) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Change in physical functioning through the dynamic visual acuity (DVA) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Change in physical functioning through the modified clinical test of sensory interaction on balance (mCTSIB) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months
Change in physical functioning through the dynamic gait index (DGI) | 3 months
  Measured by comparing the test score change from baseline to follow up at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Tartaglia, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No